CLINICAL TRIAL: NCT04017806
Title: Study Protocol for a Prospective Observational Study Investigating the Role of Luminal Pressure on Arteriovenous Fistula Maturation
Brief Title: Investigating the Role of Luminal Pressure on Arteriovenous Fistula Maturation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201801091
Record Dates: First submitted 2019-04-23; First posted 2019-07-12 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2018-09

CONDITIONS: Arteriovenous Fistula
Keywords: arteriovenous fistula maturation; End stage renal disease; luminal pressure
MeSH Terms: conditions — Arteriovenous Fistula; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction Arteriovenous fistula (AVF) is the preferred hemodialysis vascular access due to its higher patency and lower infection rate. However, its major weakness is suboptimal maturation rate. Although that substantial risk factors for AVF maturation failure have been disclosed, a modifiable risk factor remains absent. While contemporary theory for AVF maturation failure focuses on disturbed wall shear stress, complicate assumtions and measurement preclude its clinical applicability. In the process of AVF maturation, elevated luminal pressure is required for outward remodeling, however, exccessively high luminal pressure may also be ditremental to AVF maturation, which remains to be defined. This study hypothesize that higher AVF luminal pressure is harmful to its maturation and investigate its potential as a modifiable factor to improve AVF maturation.

Methods and analysis This prospective study includes patients receiving surgical creation of native AVF. The exclusion criteria include age <20 years, inability to sign inform consent and failure to create native AVF deu to technical difficulty. Demographic and labboratory profile will be collected before AVF surgery. Vascular sonography will be performed within 1 week of AVF creation to measure the blood flow rates and diameters of AVF and its branched veins. The pressure gredient within AVF will be estimated from blood flow rates by Modified Bernoulli Equation. The primary outcome was spontaneous AVF maturation defined as provision of sufficient blood flow for hemodialysis within 2 months of its creation without any interventional procedures. The secondary outcome is assisted AVF mature, which is defined as AVF maturation within 2 months from its creation, which is aided by any interventional procedure before successful use of AVF.

Ethics and dissemination This study has been approved by the ethics committee and Institutional Review Board of Taipei Medical University.

Strengths and limitations

1. The strength of the present study is the prospective design that allows complete collection of parameters and outcomes.
2. The predictor of interest for AVF maturation is luminal pressure of AVF.
3. The study assesses hemodynamic parameters of AVF and its branched veins, including diameters, flow rates, and flow volume.
4. The luminal pressure of AVF will be estimated using Modified Bernoulli Equation.
5. The primary outcome of the study is spontaneous AVF maturation.

DETAILED DESCRIPTION:
Background: AVF is the preferred vascular access for maintenance hemodialysis. However, AVF is not an ideal vascular access without any drawback. Previous studies had revealed several risk factors of AVF maturation failure, including anemia, diabetes mellitus, and smoking. On the other hand, basic studies have revealed molecular pathogenic factors of AVF maturation failure, including localized inflammation, hypoxic injury, oscillating wall shear stress, uremic milieu and oxidative stress. Despite of these substantial studies exploring the role of pathogenic factors, a modifiable pathogenic factor that is applicable to improve AVF maturation remains lacking.

Maturation failure of AVF results from luminal stenosis due to neointimal hyperplasia, signifying thickening of subintimal area caused by proliferation of myofibroblast, which is remarkably stained for α-smooth muscle actin and vimentin. Neointimal hyperplasia of AVF occurs mainly at the arteriovenous junction and venous limb of AVF, where venous endothelium is exposed to non-physiologically high blood flow rate, oscillatory shear stress and pulsatile stretching strain by arterial blood flow, suggesting the role of altered hemodynamics on AVF subintimal proliferation. It has also been reported that endothelial cells from arterial and venous parts of circulation system show different genetic expression, indicating that different hemodynamic environment regulates phenotypes of endothelial cells. Therefore, it is reasonable that elevated luminal pressure may stimulate proliferation in venous endothelium of AVF and result in maturation failure. In contrast, elevated AVF luminal pressure also provides stretching force for outward remodeling, which is required for AVF maturation. Therefore, this prospective observational study is conducted to investigate the optimal AVF luminal pressure for AVF maturation, which may be modified surgically or pharmaceutically to improve AVF maturation rate.

Specific aims Aim 1: To characterize the altered blood flow rates and luminal pressures in different segments of AVF. Aim 2: To characterize the association between luminal pressures and vessel diameters of different segments of AVF. Aim 3: To investigate the association between AVF luminal pressure and AVF maturation rate. Aim 4: To investigate the association between AVF luminal pressure and known risk factors of AVF maturation failure.

Methods and analysis: This prospective observational study is mainly aimed to investigate the association between AVF luminal pressure and maturation rate. Patients who meet the following eligibility criteria are eligible for enrollment: (1) Patient at pre-dialysis or post-dialysis status who undergoes surgical creation of native AVF for hemodialysis will be included. (2) AVF created at both radial and brachial arteries are eligible for inclusion. Exclusion criteria: (1) Patients at age <20 years old will be excluded (2) Patients who are unconscious or unable to sign the inform consent will be excluded (3) Patient in whom native AVF creation is shifted to arteriovenous graft placement due to technical difficulty will be excluded from this study. The recruit of participants, collection of parameters, and confirmation of the outcomes are performed by a full-time study nurse.

Statistic methods: Continuous variables will be expressed as mean ± standard deviation, while nominal variables are expressed in frequency and percentage. Comparisons of continuous variables will be performed using the two-tailed t-test for unpaired samples or Welch's t-test as appropriate. Comparisons of nominal variables will be performed using the Chi-square test or Fisher's exact test as appropriate. Multivariate logistic regression test will be used to evaluate the association between predictor variables and outcome variables. Statistical significance will be defined by a P value of <0.05. The statistics will be performed using SAS 9.4 (SAS Institute Inc, Cary, NC, USA). G*Power 3.1.9.4 was used to estimate the sample size to reach statistical significance in the t-test. Assuming the effect size to be 0.6. Under the condition that α error is defined as 0.05; power was defined as 0.8; and the allocation ratio was defined as 1. Therefore, the sample size required to achieve statistical significance is 90 patients. The data used for the study will be preserved and analyzed by the primary investigator. The data is accessible only to the primary investigator and study nurse for data safety. The data will be preserved for 2 years after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hemodialysis who receiving AVF.
2. AVF created at both radial and brachial arteries

Exclusion Criteria:

1. Patients at age <20 years old
2. Patients who are unconscious or unable to sign the inform consent
3. Patient in whom native AVF creation is shifted to arteriovenous graft placement

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who receives surgical anastomosis of hemodialysis AVF will be included, whether the patient is a pre-dialysis patient, fresh uremic patient or who already on dialysis treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-05-07 (Estimated); Study Completion 2020-05-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is spontaneous AVF maturation. | 2 months
  Spontaneous AVF maturation, which is defined as successful AVF puncture in hemodialysis for 6 consecutive sessions without any interventional procedure within 2 months.

SECONDARY OUTCOMES:
The secondary outcome is assisted AVF mature. | 2 months
  Assisted AVF maturation, which is defined as successful AVF puncture in hemodialysis for 6 consecutive sessions with any interventional procedure within 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-te Liu, MD, Study Director — Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan
Locations (1):
- Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bo S, Cavallo-Perin P, Gentile L, Repetti E, Pagano G. Hypouricemia and hyperuricemia in type 2 diabetes: two different phenotypes. Eur J Clin Invest. 2001 Apr;31(4):318-21. doi: 10.1046/j.1365-2362.2001.00812.x. PMID 11298778
- [Background] Edvardsson VO, Kaiser BA, Polinsky MS, Palmer JA, Quien R, Baluarte HJ. Natural history and etiology of hyperuricemia following pediatric renal transplantation. Pediatr Nephrol. 1995 Feb;9(1):57-60. doi: 10.1007/BF00858973. PMID 7742224
- [Background] Chonchol M, Shlipak MG, Katz R, Sarnak MJ, Newman AB, Siscovick DS, Kestenbaum B, Carney JK, Fried LF. Relationship of uric acid with progression of kidney disease. Am J Kidney Dis. 2007 Aug;50(2):239-47. doi: 10.1053/j.ajkd.2007.05.013. PMID 17660025
- [Background] Bellomo G, Venanzi S, Verdura C, Saronio P, Esposito A, Timio M. Association of uric acid with change in kidney function in healthy normotensive individuals. Am J Kidney Dis. 2010 Aug;56(2):264-72. doi: 10.1053/j.ajkd.2010.01.019. Epub 2010 Apr 10. PMID 20385436
- [Background] Sonoda H, Takase H, Dohi Y, Kimura G. Uric acid levels predict future development of chronic kidney disease. Am J Nephrol. 2011;33(4):352-7. doi: 10.1159/000326848. Epub 2011 Mar 25. PMID 21430373
- [Background] Iseki K, Oshiro S, Tozawa M, Iseki C, Ikemiya Y, Takishita S. Significance of hyperuricemia on the early detection of renal failure in a cohort of screened subjects. Hypertens Res. 2001 Nov;24(6):691-7. doi: 10.1291/hypres.24.691. PMID 11768729
- [Background] Kang DH, Nakagawa T, Feng L, Watanabe S, Han L, Mazzali M, Truong L, Harris R, Johnson RJ. A role for uric acid in the progression of renal disease. J Am Soc Nephrol. 2002 Dec;13(12):2888-97. doi: 10.1097/01.asn.0000034910.58454.fd. PMID 12444207
- [Background] Anker SD, Doehner W, Rauchhaus M, Sharma R, Francis D, Knosalla C, Davos CH, Cicoira M, Shamim W, Kemp M, Segal R, Osterziel KJ, Leyva F, Hetzer R, Ponikowski P, Coats AJ. Uric acid and survival in chronic heart failure: validation and application in metabolic, functional, and hemodynamic staging. Circulation. 2003 Apr 22;107(15):1991-7. doi: 10.1161/01.CIR.0000065637.10517.A0. Epub 2003 Apr 21. PMID 12707250
- [Background] Hsu SP, Pai MF, Peng YS, Chiang CK, Ho TI, Hung KY. Serum uric acid levels show a 'J-shaped' association with all-cause mortality in haemodialysis patients. Nephrol Dial Transplant. 2004 Feb;19(2):457-62. doi: 10.1093/ndt/gfg563. PMID 14736974
- [Background] Suliman ME, Johnson RJ, Garcia-Lopez E, Qureshi AR, Molinaei H, Carrero JJ, Heimburger O, Barany P, Axelsson J, Lindholm B, Stenvinkel P. J-shaped mortality relationship for uric acid in CKD. Am J Kidney Dis. 2006 Nov;48(5):761-71. doi: 10.1053/j.ajkd.2006.08.019. PMID 17059995
- [Background] Siu YP, Leung KT, Tong MK, Kwan TH. Use of allopurinol in slowing the progression of renal disease through its ability to lower serum uric acid level. Am J Kidney Dis. 2006 Jan;47(1):51-9. doi: 10.1053/j.ajkd.2005.10.006. PMID 16377385
- [Background] Goicoechea M, de Vinuesa SG, Verdalles U, Ruiz-Caro C, Ampuero J, Rincon A, Arroyo D, Luno J. Effect of allopurinol in chronic kidney disease progression and cardiovascular risk. Clin J Am Soc Nephrol. 2010 Aug;5(8):1388-93. doi: 10.2215/CJN.01580210. Epub 2010 Jun 10. PMID 20538833
- [Background] Wang H, Wei Y, Kong X, Xu D. Effects of urate-lowering therapy in hyperuricemia on slowing the progression of renal function: a meta-analysis. J Ren Nutr. 2013 Sep;23(5):389-96. doi: 10.1053/j.jrn.2012.08.005. Epub 2012 Nov 4. PMID 23131573
- [Background] Levy G, Cheetham TC. Is It Time to Start Treating Asymptomatic Hyperuricemia? Am J Kidney Dis. 2015 Dec;66(6):933-5. doi: 10.1053/j.ajkd.2015.09.002. No abstract available. PMID 26593311
- [Background] Hande KR, Noone RM, Stone WJ. Severe allopurinol toxicity. Description and guidelines for prevention in patients with renal insufficiency. Am J Med. 1984 Jan;76(1):47-56. doi: 10.1016/0002-9343(84)90743-5. PMID 6691361
- [Background] Kamatani N, Fujimori S, Hada T, Hosoya T, Kohri K, Nakamura T, Ueda T, Yamamoto T, Yamanaka H, Matsuzawa Y. An allopurinol-controlled, multicenter, randomized, open-label, parallel between-group, comparative study of febuxostat (TMX-67), a non-purine-selective inhibitor of xanthine oxidase, in patients with hyperuricemia including those with gout in Japan: phase 2 exploratory clinical study. J Clin Rheumatol. 2011 Jun;17(4 Suppl 2):S44-9. doi: 10.1097/RHU.0b013e31821d352f. PMID 21654269
- [Background] Tanaka K, Nakayama M, Kanno M, Kimura H, Watanabe K, Tani Y, Hayashi Y, Asahi K, Terawaki H, Watanabe T. Renoprotective effects of febuxostat in hyperuricemic patients with chronic kidney disease: a parallel-group, randomized, controlled trial. Clin Exp Nephrol. 2015 Dec;19(6):1044-53. doi: 10.1007/s10157-015-1095-1. Epub 2015 Feb 13. PMID 25676011
- [Background] Sircar D, Chatterjee S, Waikhom R, Golay V, Raychaudhury A, Chatterjee S, Pandey R. Efficacy of Febuxostat for Slowing the GFR Decline in Patients With CKD and Asymptomatic Hyperuricemia: A 6-Month, Double-Blind, Randomized, Placebo-Controlled Trial. Am J Kidney Dis. 2015 Dec;66(6):945-50. doi: 10.1053/j.ajkd.2015.05.017. Epub 2015 Jul 30. PMID 26233732
- [Result] Madero M, Sarnak MJ, Wang X, Greene T, Beck GJ, Kusek JW, Collins AJ, Levey AS, Menon V. Uric acid and long-term outcomes in CKD. Am J Kidney Dis. 2009 May;53(5):796-803. doi: 10.1053/j.ajkd.2008.12.021. Epub 2009 Mar 20. PMID 19303683
- [Derived] Cheng HS, Chang TI, Chen CH, Hsu SC, Hsieh HL, Chen CY, Huang WC, Sue YM, Lin FY, Shih CM, Chen JW, Lin SJ, Huang PH, Liu CT. Study protocol for a prospective observational study to investigate the role of luminal pressure on arteriovenous fistula maturation. Medicine (Baltimore). 2019 Oct;98(40):e17238. doi: 10.1097/MD.0000000000017238. PMID 31577715